CLINICAL TRIAL: NCT02873221
Title: A Multicenter, Randomized, Open-Label Extension Study to Evaluate the Long-Term Safety and Tolerability of Oral Ubrogepant in the Acute Treatment of Migraine With or Without Aura
Brief Title: An Extension Study to Evaluate the Long-Term Safety and Tolerability of Ubrogepant in the Treatment of Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBR-MD-04
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Migraine, With or Without Aura
MeSH Terms: conditions — Migraine Disorders | interventions — ubrogepant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Usual Care (Active Comparator): Usual Care as prescribed by the physician as standard of care in clinical practice for the treatment of migraine attacks for up to 1 year.
  Interventions: Drug: Usual Care
- Ubrogepant 50 mg (Experimental): Ubrogepant 50 mg tablet orally plus placebo-matching ubrogepant tablet for the treatment of a qualifying migraine attack for up to 8 treatments every 4 weeks for up to 1 year. Participants may choose to take a second dose orally after the initial dose if migraine continues or returns.
  Interventions: Drug: Ubrogepant; Drug: Placebo-matching Ubrogepant
- Ubrogepant 100 mg (Experimental): Ubrogepant 100 mg (two 50 mg tablets) orally for the treatment of a qualifying migraine attack for up to 8 treatments every 4 weeks for up to 1 year. Participants may choose to take a second dose orally after the initial dose if migraine continues or returns.
  Interventions: Drug: Ubrogepant

INTERVENTIONS:
Drug: Ubrogepant — Ubrogepant tablet(s) orally for the treatment of a qualifying migraine attack.
  Arms: Ubrogepant 100 mg; Ubrogepant 50 mg
Drug: Placebo-matching Ubrogepant — Ubrogepant placebo-matching tablet orally for the treatment of a qualifying migraine attack.
  Arms: Ubrogepant 50 mg
Drug: Usual Care — Treatment for a migraine as prescribed by the physician as standard of care in clinical practice.
  Arms: Usual Care

SUMMARY:
This study will evaluate the long-term safety and tolerability of intermittent treatment with ubrogepant for the acute treatment of migraine over 1 year.

DETAILED DESCRIPTION:
Usual care is the open-label control arm. Dose of ubrogepant (50 mg or 100 mg) will be double-blind for active treatment arms.

ELIGIBILITY:
Inclusion Criteria:

-Completed study UBR-MD-01(NCT02828020) or UBR-MD-02(NCT02867709).

Exclusion Criteria:

* Patients with clinically significant electrocardiogram (ECG), vital sign, physical exam, or laboratory abnormalities
* Requirement for a medication during the study that is on the list of prohibited medications.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1254 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adele Thorpe, Study Director — Allergan
Locations (177):
- United States (177):
  - Radiant Research, Inc., Birmingham, Alabama
  - East Family Physicians PC/Radiant Research, Inc., Chandler, Arizona
  - Desert Clinical Research /Radiant Research, Inc., Mesa, Arizona
  - Xenoscience, Inc., Phoenix, Arizona
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Radiant Research Inc., Tucson, Arizona
  - Orange Grove Family Practice/Radiant Research, Inc., Tucson, Arizona
  - Principals Research Group, Inc., Hot Springs, Arkansas
  - Arkansas Clinical Research, Little Rock, Arkansas
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Axiom Research, Apple Valley, California
  - Hope Clinical Research, Canoga Park, California
  - Med Center Medical Clinic Carmichael, Carmichael, California
  - Axiom Research, LLC, Colton, California
  - Pharmacology Research Institute, Encino, California
  - Encino Research Center/T Joseph Raoof MD Inc, Encino, California
  - Neuro-Pain Medical Center, Inc, Fresno, California
  - California Headache and Balance Center, Fresno, California
  - Neurology Center of North Orange County, Fullerton, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Sun Valley Research Center, Imperial, California
  - Grossmont Center For Clinical Research, La Mesa, California
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pacific Institute of Medical Research, Los Angeles, California
  - Synergy San Diego, National City, California
  - Pharmacology Research Institute, Newport Beach, California
  - Newport Beach Clinical Research Associates, Inc., Newport Beach, California
  - Rancho Cucamonga Clinical Research, Rancho Cucamonga, California
  - Desert Valley Research, Rancho Mirage, California
  - George J Rederich MD, Inc., Redondo Beach, California
  - Artemis Institute For Clinical Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Southern California Research Center, Simi Valley, California
  - Encompass Clinical Research, Spring Valley, California
  - Radiant Research, Vista, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Clinicos LLC, Colorado Springs, Colorado
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Delta Waves, Inc, Colorado Springs, Colorado
  - Denver Neurological Research, Denver, Colorado
  - Summit Headache and Neurologic Institute, Englewood, Colorado
  - Advanced Neurosciences Research, Fort Collins, Colorado
  - Associated Neurologists, PC, Danbury, Connecticut
  - Associated Neurologists of Southern Connecticut, PC, Fairfield, Connecticut
  - Aventura Neurological Associates, PA, Aventura, Florida
  - Clinical Research South Florida, Coral Gables, Florida
  - Avail Clinical Research, DeLand, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Wilks & Safirstein MD PA D/B/A MD Clinical, Hallandale, Florida
  - Infinity Clinical Research, Hollywood, Florida
  - Broward Research, Hollywood, Florida
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Neurology Associates, P.A., Maitland, Florida
  - LCC Medical Research, Miami, Florida
  - Well Pharma Medical Research, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Clinical Neuroscience Solutions, Inc - Memphis, TN, Orlando, Florida
  - Palm Beach Neurological Center / Advanced Research Consultants, Inc., Palm Beach Gardens, Florida
  - Qps Mra, Llc, South Miami, Florida
  - Meridien Research, Spring Hill, Florida
  - University of South Florida, Tampa, Florida
  - Meridien Research, Tampa, Florida
  - Neurology Research Institute Palm Beach, West Palm Beach, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Midtown Neurology, Atlanta, Georgia
  - NeuroTrials Research Inc, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Michigan Ave. Internists /Radiant Research, Inc., Chicago, Illinois
  - Cedar Crosse Research Center, Chicago, Illinois
  - Great Lakes Clinical Trials, LLC, Chicago, Illinois
  - Robbins Headache Clinic, Riverwoods, Illinois
  - Deaconess Clinic Inc., Evansville, Indiana
  - Josephson Wallack Munshower Neurology, P.C., Indianapolis, Indiana
  - Rowe Neurology Institute, Lenexa, Kansas
  - College Park Family Care Center Physicians Group- Neurology Research Dept, Overland Park, Kansas
  - Kansas Institute of Research, Overland Park, Kansas
  - Kentucky Pediatric Research Inc, Bardstown, Kentucky
  - Norton Neurology Services, Louisville, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Pharma Site Research, Baltimore, Maryland
  - Seton Medical Group, Baltimore, Maryland
  - Boston Clinical Trials Inc, Boston, Massachusetts
  - BTC of New Bedford, New Bedford, Massachusetts
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - Beacon Clinical Research, LLC, Quincy, Massachusetts
  - Medvadis Research Corporation, Watertown, Massachusetts
  - New England Regional Headache Center, Worcester, Massachusetts
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - Quest Research Institute, Farmington Hills, Michigan
  - Women's Health Care Specialists, Kalamazoo, Michigan
  - The Minneapolis Clinic of Neurology, Ltd., Golden Valley, Minnesota
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - The Headache Center, Ridgeland, Mississippi
  - Clinvest, Springfield, Missouri
  - Prairie Fields Family Medicine, Fremont, Nebraska
  - Clinical Research Advantage, Inc/Synexus USA, Omaha, Nebraska
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Diagnostic Center of Medicine - Durango / Radiant Research, Inc., Las Vegas, Nevada
  - Princeton Medical Institute, Princeton, New Jersey
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - DENT Neurosciences Research Center, Amherst, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - Central New York Clinical Research, Manlius, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Headache Wellness Center, Greensboro, North Carolina
  - Neurology Associates, P.A., Hickory, North Carolina
  - Lake Shore Clinical Research, LLC, Mooresville, North Carolina
  - Wake Research Associates LLC, Raleigh, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Plains Clinical Research Center, LLC, Fargo, North Dakota
  - Radiant Research, Inc., Akron, Ohio
  - Neuro-Behavioral Clinical Research, Inc, Canton, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Sentral Clinical Research Services, Cincinnati, Ohio
  - Patient Priority Clinical Sites, Cincinnati, Ohio
  - University of cincinnati, Cincinnati, Ohio
  - CTI Clinical research Center, Cincinnati, Ohio
  - Radiant Research, Inc, Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Ohio Clinical Research, LLC, Cleveland, Ohio
  - Aventiv Research Inc., Columbus, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - NPC Research, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Sooner Clinical Research Inc, Oklahoma City, Oklahoma
  - Summit Research Network Inc., Portland, Oregon
  - Oregon Center For Clinical Investigations Inc, Portland, Oregon
  - Clinical Research Philadelphia, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Lincoln Research, Lincoln, Rhode Island
  - Radiant Research, Anderson, South Carolina
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Vista Clinical Research, Columbia, South Carolina
  - Hillcrest Clinical Research LLC, Simpsonville, South Carolina
  - Clinsearch, LLC, Chattanooga, Tennessee
  - Middle Tennessee Clinical Research, Fayetteville, Tennessee
  - Holston Medical Group, P.C., Kingsport, Tennessee
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - CNS Healthcare, Memphis, Tennessee
  - Future Search Trials, Austin, Texas
  - Tekton Research, Austin, Texas
  - Texas Neurology, P.A., Dallas, Texas
  - Futuresearch Trials of Dallas, LP, Dallas, Texas
  - Radiant Research, Inc., Dallas, Texas
  - Research Trials Worldwide, LLC, Humble, Texas
  - Red Star Research, LLC, Lake Jackson, Texas
  - Clinical Trials Texas, Inc, San Antonio, Texas
  - Road Runner Research, San Antonio, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic Draper, Draper, Utah
  - Advanced Research Institute, Ogden, Utah
  - Granger Medical Clinic - Riverton, Riverton, Utah
  - Optimum Clinical Research, Inc., Salt Lake City, Utah
  - Highland Clinical Reserach, Salt Lake City, Utah
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Clinical Research Associates Tidewater, Norfolk, Virginia
  - Blue Ridge Research Center, Roanoke, Virginia
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Sentara Neurology Specialists, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - The Polyclinic, Seattle, Washington
  - South Puget Sound Neurology, Tacoma, Washington
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- [Derived] Lipton RB, Dodick DW, Goadsby PJ, Burstein R, Adams AM, Lai J, Yu SY, Finnegan M, Kuang AW, Trugman JM. Efficacy of Ubrogepant in the Acute Treatment of Migraine With Mild Pain vs Moderate or Severe Pain. Neurology. 2022 Oct 25;99(17):e1905-e1915. doi: 10.1212/WNL.0000000000201031. Epub 2022 Aug 17. PMID 35977836
- [Derived] Blumenfeld AM, Knievel K, Manack Adams A, Severt L, Butler M, Lai H, Dodick DW. Ubrogepant Is Safe and Efficacious in Participants Taking Concomitant Preventive Medication for Migraine: A Pooled Analysis of Phase 3 Trials. Adv Ther. 2022 Jan;39(1):692-705. doi: 10.1007/s12325-021-01923-3. Epub 2021 Dec 7. PMID 34874514
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period
Arm/Group | Usual Care | Ubrogepant 50 mg | Ubrogepant 100 mg
Started | 417 | 417 | 420
Safety Population: Received Study Drug | 417 | 404 | 409
Completed | 329 | 291 | 315
Not Completed | 88 | 126 | 105
Not completed — Other Miscellaneous Reasons | 0 | 2 | 1
Not completed — Non-Compliance with Study Drug | 0 | 3 | 2
Not completed — Protocol Violation | 2 | 5 | 8
Not completed — Pregnancy | 4 | 6 | 3
Not completed — Lack of Qualifying Event | 0 | 3 | 1
Not completed — Withdrawal of Consent | 52 | 51 | 41
Not completed — Lack of Efficacy | 0 | 17 | 12
Not completed — Adverse Event | 4 | 9 | 11
Not completed — Lost to Follow-up | 26 | 30 | 26
Period: Safety Follow-up Period
Arm/Group | Usual Care | Ubrogepant 50 mg | Ubrogepant 100 mg
Started | 350 | 356 | 364
Completed | 343 | 339 | 350
Not Completed | 7 | 17 | 14
Not completed — Other Miscellaneous Reasons | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Lost to Follow-up | 3 | 5 | 5
Not completed — Withdrawal of Consent | 4 | 10 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Ubrogepant 50 mg | Ubrogepant 100 mg | Total
Number analyzed (Participants) | 417 | 417 | 420 | 1254
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.7 (11.7) | 42.2 (12.2) | 41.2 (11.2) | 41.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 367 | 384 | 375 | 1126
  Male | 50 | 33 | 45 | 128
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 356 | 358 | 345 | 1059
  Black or African American | 50 | 52 | 61 | 163
  Asian | 3 | 2 | 5 | 10
  American Indian or Alaska Native | 4 | 2 | 3 | 9
  Native Hawaiian/Other Pacific Islander | 0 | 1 | 2 | 3
  Multiple | 4 | 2 | 4 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 62 | 64 | 59 | 185
  Not Hispanic or Latino | 355 | 353 | 361 | 1069

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1 Treatment Emergent Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAEs are AEs with an onset that occurs after receiving study drug.
Time Frame: 56 Weeks
Population: The Safety population is defined separately below for the ubrogepant arms and the usual-care arm.
  Ubrogepant arms: All randomized patients who received ≥ 1 dose of treatment. Usual care arm: All randomized patients in the usual-care arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Usual Care | Ubrogepant 50 mg | Ubrogepant 100 mg
Number analyzed (Participants) | 417 | 404 | 409
Percentage of Participants | 65 | 66.3 | 72.6

2. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Values
Description: Hematology, Chemistry and Urinalysis results considered potentially clinically significant (PCS) meeting either the lower-limit or higher-limit PCS criteria.
Time Frame: 56 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Ubrogepant 50 mg | Ubrogepant 100 mg
Number analyzed (Participants) | 417 | 404 | 409
Participants
  Basophils Absolute Cell Count (10**9/L) >2×ULN: number analyzed (Participants) | 397 | 397 | 405
  Basophils Absolute Cell Count (10**9/L) >2×ULN | 0 | 0 | 0
  Eosinophils Absolute Cell Count (10**9/L) >2×ULN: number analyzed (Participants) | 397 | 397 | 405
  Eosinophils Absolute Cell Count (10**9/L) >2×ULN | 1 | 0 | 1
  Hematocrit (RATIO) <0.9×LLN: number analyzed (Participants) | 397 | 396 | 406
  Hematocrit (RATIO) <0.9×LLN | 3 | 2 | 6
  Hematocrit (RATIO) >1.1×ULN: number analyzed (Participants) | 397 | 396 | 406
  Hematocrit (RATIO) >1.1×ULN | 2 | 0 | 1
  Hemoglobin (g/L) <0.9×LLN: number analyzed (Participants) | 395 | 395 | 405
  Hemoglobin (g/L) <0.9×LLN | 7 | 3 | 6
  Hemoglobin (g/L) >1.1×ULN: number analyzed (Participants) | 395 | 395 | 405
  Hemoglobin (g/L) >1.1×ULN | 2 | 0 | 1
  Lymphocytes Absolute Cell Count (10**9/L) <0.7×LLN: number analyzed (Participants) | 395 | 397 | 404
  Lymphocytes Absolute Cell Count (10**9/L) <0.7×LLN | 11 | 5 | 5
  Lymphocytes Absolute Cell Count (10**9/L) >1.3×ULN: number analyzed (Participants) | 395 | 397 | 404
  Lymphocytes Absolute Cell Count (10**9/L) >1.3×ULN | 8 | 6 | 8
  Monocytes Absolute Cell Count (10**9/L) <0.5×LLN: number analyzed (Participants) | 397 | 397 | 405
  Monocytes Absolute Cell Count (10**9/L) <0.5×LLN | 0 | 0 | 0
  Monocytes Absolute Cell Count (10**9/L) >2×ULN: number analyzed (Participants) | 397 | 397 | 405
  Monocytes Absolute Cell Count (10**9/L) >2×ULN | 0 | 0 | 0
  Neutrophils Absolute Cell Count (10**9/L) <0.7×LLN: number analyzed (Participants) | 396 | 395 | 401
  Neutrophils Absolute Cell Count (10**9/L) <0.7×LLN | 6 | 5 | 6
  Neutrophils Absolute Cell Count (10**9/L) >1.3×ULN: number analyzed (Participants) | 396 | 395 | 401
  Neutrophils Absolute Cell Count (10**9/L) >1.3×ULN | 22 | 14 | 17
  Platelet Count (Thrombocytes) (10**9/L) <0.5×LLN: number analyzed (Participants) | 394 | 394 | 404
  Platelet Count (Thrombocytes) (10**9/L) <0.5×LLN | 0 | 0 | 0
  Platelet Count (Thrombocytes) (10**9/L) >1.5×ULN: number analyzed (Participants) | 394 | 394 | 404
  Platelet Count (Thrombocytes) (10**9/L) >1.5×ULN | 2 | 2 | 1
  Red Blood Cell Count (10**12/L) <0.9×LLN: number analyzed (Participants) | 395 | 398 | 401
  Red Blood Cell Count (10**12/L) <0.9×LLN | 1 | 5 | 3
  Red Blood Cell Count (10**12/L) >1.1×ULN: number analyzed (Participants) | 395 | 398 | 401
  Red Blood Cell Count (10**12/L) >1.1×ULN | 2 | 2 | 2
  White Blood Cell Count (10**9/L) <0.9×LLN: number analyzed (Participants) | 396 | 397 | 403
  White Blood Cell Count (10**9/L) <0.9×LLN | 17 | 9 | 17
  White Blood Cell Count (10**9/L) >1.5×ULN: number analyzed (Participants) | 396 | 397 | 403
  White Blood Cell Count (10**9/L) >1.5×ULN | 5 | 2 | 4
  Alanine Aminotransferase (SGPT) (U/L) >3×ULN: number analyzed (Participants) | 397 | 399 | 406
  Alanine Aminotransferase (SGPT) (U/L) >3×ULN | 4 | 4 | 8
  Albumin (g/L) <0.8×LLN: number analyzed (Participants) | 397 | 399 | 406
  Albumin (g/L) <0.8×LLN | 0 | 1 | 0
  Albumin (g/L) >1.2×ULN: number analyzed (Participants) | 397 | 399 | 406
  Albumin (g/L) >1.2×ULN | 0 | 0 | 0
  Alkaline Phosphatase (U/L) >3×ULN: number analyzed (Participants) | 396 | 399 | 406
  Alkaline Phosphatase (U/L) >3×ULN | 0 | 0 | 0
  Aspartate Aminotransferase (SGOT) (U/L) >3×ULN: number analyzed (Participants) | 397 | 399 | 406
  Aspartate Aminotransferase (SGOT) (U/L) >3×ULN | 2 | 2 | 9
  Bicarbonate (HCO3) (mmol/L) <0.9×LLN: number analyzed (Participants) | 386 | 392 | 395
  Bicarbonate (HCO3) (mmol/L) <0.9×LLN | 25 | 22 | 37
  Bicarbonate (HCO3) (mmol/L) >1.1×ULN: number analyzed (Participants) | 386 | 392 | 395
  Bicarbonate (HCO3) (mmol/L) >1.1×ULN | 0 | 0 | 0
  Bilirubin, Total (umol/L) >1.5×ULN: number analyzed (Participants) | 396 | 398 | 405
  Bilirubin, Total (umol/L) >1.5×ULN | 3 | 4 | 2
  Blood Urea Nitrogen (mmol/L) >1.5×ULN: number analyzed (Participants) | 397 | 399 | 406
  Blood Urea Nitrogen (mmol/L) >1.5×ULN | 6 | 3 | 1
  Calcium (mmol/L) <0.9×LLN: number analyzed (Participants) | 396 | 399 | 406
  Calcium (mmol/L) <0.9×LLN | 2 | 1 | 3
  Calcium (mmol/L) >1.1×ULN: number analyzed (Participants) | 396 | 399 | 406
  Calcium (mmol/L) >1.1×ULN | 0 | 0 | 0
  Chloride (mmol/L) <0.9×LLN: number analyzed (Participants) | 396 | 399 | 405
  Chloride (mmol/L) <0.9×LLN | 0 | 0 | 1
  Chloride (mmol/L) >1.1×UL: number analyzed (Participants) | 396 | 399 | 405
  Chloride (mmol/L) >1.1×UL | 0 | 0 | 0
  Cholesterol, Total (mmol/L) >1.6×ULN: number analyzed (Participants) | 397 | 397 | 405
  Cholesterol, Total (mmol/L) >1.6×ULN | 4 | 1 | 2
  Creatine Kinase (U/L) >2×ULN: number analyzed (Participants) | 392 | 395 | 398
  Creatine Kinase (U/L) >2×ULN | 56 | 43 | 57
  Creatinine (umol/L) >1.5×ULN: number analyzed (Participants) | 397 | 399 | 406
  Creatinine (umol/L) >1.5×ULN | 1 | 1 | 1
  Glucose, Non-fasting (mmol/L) <0.8×LLN: number analyzed (Participants) | 397 | 399 | 406
  Glucose, Non-fasting (mmol/L) <0.8×LLN | 0 | 0 | 0
  Glucose, Non-fasting (mmol/L) >2×ULN: number analyzed (Participants) | 397 | 399 | 406
  Glucose, Non-fasting (mmol/L) >2×ULN | 1 | 1 | 1
  Lactate Dehydrogenase (U/L) >3×ULN: number analyzed (Participants) | 397 | 399 | 406
  Lactate Dehydrogenase (U/L) >3×ULN | 0 | 0 | 0
  Phosphorus (mmol/L) <0.9×LLN: number analyzed (Participants) | 389 | 392 | 403
  Phosphorus (mmol/L) <0.9×LLN | 45 | 38 | 42
  Phosphorus (mmol/L) >1.1×ULN: number analyzed (Participants) | 389 | 392 | 403
  Phosphorus (mmol/L) >1.1×ULN | 21 | 15 | 21
  Potassium (mmol/L) <0.9×LLN: number analyzed (Participants) | 395 | 398 | 402
  Potassium (mmol/L) <0.9×LLN | 0 | 1 | 3
  Potassium (mmol/L) >1.1×ULN: number analyzed (Participants) | 395 | 398 | 402
  Potassium (mmol/L) >1.1×ULN | 28 | 32 | 33
  Protein, Total (g/L) <0.9×LLN: number analyzed (Participants) | 396 | 398 | 406
  Protein, Total (g/L) <0.9×LLN | 3 | 2 | 4
  Protein, Total (g/L) >1.1×ULN: number analyzed (Participants) | 396 | 398 | 406
  Protein, Total (g/L) >1.1×ULN | 0 | 0 | 0
  Sodium (mmol/L) <0.9×LLN: number analyzed (Participants) | 397 | 399 | 406
  Sodium (mmol/L) <0.9×LLN | 0 | 0 | 0
  Sodium (mmol/L) >1.1×ULN: number analyzed (Participants) | 397 | 399 | 406
  Sodium (mmol/L) >1.1×ULN | 0 | 0 | 2
  Triglycerides (mmol/L) >2×ULN: number analyzed (Participants) | 391 | 397 | 398
  Triglycerides (mmol/L) >2×ULN | 30 | 20 | 17
  Uric Acid (Urate) (umol/L) >1.2×ULN: number analyzed (Participants) | 390 | 392 | 406
  Uric Acid (Urate) (umol/L) >1.2×ULN | 26 | 27 | 22
  Glucose Positive: number analyzed (Participants) | 388 | 393 | 401
  Glucose Positive | 21 | 17 | 23
  pH (pH) <0.9×LLN: number analyzed (Participants) | 397 | 398 | 406
  pH (pH) <0.9×LLN | 0 | 0 | 0
  pH (pH) >1.1×ULN: number analyzed (Participants) | 397 | 398 | 406
  pH (pH) >1.1×ULN | 0 | 0 | 0
  Protein (g/L) Positive: number analyzed (Participants) | 377 | 381 | 380
  Protein (g/L) Positive | 0 | 0 | 0
  Specific Gravity >1.1×ULN: number analyzed (Participants) | 397 | 399 | 406
  Specific Gravity >1.1×ULN | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiograms (ECGs) Findings
Description: ECG findings considered potentially clinically significant (PCS) meeting either the lower-limit or higher-limit PCS criteria.
Time Frame: 56 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Ubrogepant 50 mg | Ubrogepant 100 mg
Number analyzed (Participants) | 417 | 404 | 409
Participants
  PR interval (msec) PR >= 250: number analyzed (Participants) | 385 | 389 | 399
  PR interval (msec) PR >= 250 | 0 | 0 | 0
  QRS interval (msec) QRS >= 150: number analyzed (Participants) | 385 | 389 | 399
  QRS interval (msec) QRS >= 150 | 1 | 1 | 0
  QTc Bazett (msec) QTcB > 500: number analyzed (Participants) | 385 | 388 | 399
  QTc Bazett (msec) QTcB > 500 | 0 | 0 | 0
  QTc Bazett (msec) Increase > 60 (msec): number analyzed (Participants) | 385 | 388 | 399
  QTc Bazett (msec) Increase > 60 (msec) | 0 | 1 | 5
  QTc Fridericia (msec) QTcF > 500: number analyzed (Participants) | 385 | 388 | 399
  QTc Fridericia (msec) QTcF > 500 | 0 | 0 | 0
  QTc Fridericia (msec) Increase > 60 (msec): number analyzed (Participants) | 385 | 388 | 399
  QTc Fridericia (msec) Increase > 60 (msec) | 1 | 0 | 0

4. Secondary Outcome: Number of Participants With Clinically Significant Vital Sign Measurements
Description: Vital sign measurements considered potentially clinically significant (PCS) meeting either the lower-limit or higher-limit PCS criteria.
Time Frame: 56 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Ubrogepant 50 mg | Ubrogepant 100 mg
Number analyzed (Participants) | 417 | 404 | 409
Participants
  SBP (mmHg) (Sitting) <= 90 and Decrease of >= 20: number analyzed (Participants) | 398 | 400 | 406
  SBP (mmHg) (Sitting) <= 90 and Decrease of >= 20 | 11 | 20 | 12
  SBP (mmHg) (Sitting) >= 180 and Increase of >= 20: number analyzed (Participants) | 398 | 400 | 406
  SBP (mmHg) (Sitting) >= 180 and Increase of >= 20 | 0 | 0 | 1
  SBP (mmHg) (Standing) <= 90 and Decrease of >= 20: number analyzed (Participants) | 398 | 400 | 406
  SBP (mmHg) (Standing) <= 90 and Decrease of >= 20 | 12 | 11 | 11
  SBP (mmHg) (Standing) >= 180 and Increase of >= 20: number analyzed (Participants) | 398 | 400 | 406
  SBP (mmHg) (Standing) >= 180 and Increase of >= 20 | 0 | 0 | 1
  Standing - Sitting SBP (mmHg) <= -20: number analyzed (Participants) | 398 | 400 | 406
  Standing - Sitting SBP (mmHg) <= -20 | 58 | 40 | 49
  DBP (mmHg) (Sitting) <= 50 and Decrease of >= 15: number analyzed (Participants) | 398 | 400 | 406
  DBP (mmHg) (Sitting) <= 50 and Decrease of >= 15 | 6 | 5 | 4
  DBP (mmHg) (Sitting) >= 105 and Increase of >= 15: number analyzed (Participants) | 398 | 400 | 406
  DBP (mmHg) (Sitting) >= 105 and Increase of >= 15 | 6 | 3 | 6
  DBP (mmHg) (Standing) <= 50 and Decrease of >= 15: number analyzed (Participants) | 398 | 400 | 406
  DBP (mmHg) (Standing) <= 50 and Decrease of >= 15 | 5 | 4 | 4
  DBP (mmHg) (Standing) >= 105 and Increase of >= 15: number analyzed (Participants) | 398 | 400 | 406
  DBP (mmHg) (Standing) >= 105 and Increase of >= 15 | 12 | 14 | 11
  Standing - Sitting DBP (mmHg) <= -15: number analyzed (Participants) | 398 | 400 | 406
  Standing - Sitting DBP (mmHg) <= -15 | 38 | 42 | 36
  PR (beats/min) (Sitting) <= 50, Decrease of >= 15: number analyzed (Participants) | 398 | 400 | 406
  PR (beats/min) (Sitting) <= 50, Decrease of >= 15 | 4 | 5 | 7
  PR (beats/min) (Sitting) >= 120, Increase of >= 15: number analyzed (Participants) | 398 | 400 | 406
  PR (beats/min) (Sitting) >= 120, Increase of >= 15 | 1 | 2 | 1
  PR (beats/min) (Standing) <= 50, Decrease of >= 15: number analyzed (Participants) | 398 | 400 | 406
  PR (beats/min) (Standing) <= 50, Decrease of >= 15 | 2 | 3 | 3
  PR (beats/min)(Standing) >= 120, Increase of >= 15: number analyzed (Participants) | 398 | 400 | 406
  PR (beats/min)(Standing) >= 120, Increase of >= 15 | 14 | 9 | 13
  Standing - Sitting Pulse Rate (beats/min) >= 25: number analyzed (Participants) | 398 | 400 | 406
  Standing - Sitting Pulse Rate (beats/min) >= 25 | 42 | 37 | 35
  Weight (kg) Decrease of >= 7%: number analyzed (Participants) | 398 | 400 | 406
  Weight (kg) Decrease of >= 7% | 58 | 48 | 53
  Weight (kg) Increase of >= 7%: number analyzed (Participants) | 398 | 400 | 406
  Weight (kg) Increase of >= 7% | 73 | 69 | 61

5. Secondary Outcome: Number of Participants Experiencing Suicidal Ideation or Suicidal Behavior Based on Columbia-Suicide Severity Rating Scale (C-SSRS) Using 5-Point Scales
Description: On the C-SSRS, the 5 types of suicidal ideation are:
  Type 1: "Wish to be dead" Type 2: Non-specific active suicidal thoughts Type 3: "Active suicidal ideation with any methods (not plan) without intent to act" Type 4: "Active suicidal ideation with some intent to act, without specific plan" Type 5: "Active suicidal ideation with specific plan and intent"
Time Frame: 56 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Ubrogepant 50 mg | Ubrogepant 100 mg
Number analyzed (Participants) | 417 | 404 | 409
Participants
  Suicidal Ideation | 5 | 3 | 2
  Suicidal Behavior | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 56 weeks.
Description: The Safety population is defined separately below for the ubrogepant arms and the usual-care arm.
  Ubrogepant arms: All randomized patients who received ≥ 1 dose of treatment.
  Usual care arm: All randomized patients in the usual-care arm.
Arm/Group | Usual Care | Ubrogepant 50 mg | Ubrogepant 100 mg
All-Cause Mortality (participants affected / at risk) | 0/417 | 0/404 | 0/409
Serious Adverse Events (participants affected / at risk) | 17/417 | 9/404 | 12/409
Other Adverse Events (participants affected / at risk) | 132/417 | 125/404 | 138/409
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=417) | Ubrogepant 50 mg (N=404) | Ubrogepant 100 mg (N=409)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Device allergy (Immune system disorders) | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Femoral hernia incarcerated (Gastrointestinal disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Substance-induced mood disorder (Psychiatric disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=417) | Ubrogepant 50 mg (N=404) | Ubrogepant 100 mg (N=409)
Nasopharyngitis (Infections and infestations) | 33 | 33 | 47
Upper respiratory tract infection (Infections and infestations) | 48 | 47 | 44
Sinusitis (Infections and infestations) | 25 | 28 | 26
Urinary tract infection (Infections and infestations) | 23 | 22 | 26
Influenza (Infections and infestations) | 21 | 17 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT02873221/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT02873221/SAP_001.pdf